CLINICAL TRIAL: NCT03278470
Title: A Dose Block-randomized, Double Blinded, Placebo Controlled, Dose-escalation Clinical Trial to Find the Maximum Tolerable Dose After Single Oral Dose of HL237 in Healthy Male Subject
Brief Title: A Single Ascending Dose Clinical Trial to Find the Maximum Tolerable Dose of HL237 in Healthy Male Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: HL-237-101
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- HL237 50mg (Experimental): take oral tablet once
  Interventions: Drug: HL237; Drug: Placebo Oral Tablet
- HL237 100mg (Experimental): take oral tablet once
  Interventions: Drug: HL237; Drug: Placebo Oral Tablet
- HL237 200mg (Experimental): take oral tablet once
  Interventions: Drug: HL237; Drug: Placebo Oral Tablet
- HL237 400mg (Experimental): take oral tablet once
  Interventions: Drug: HL237; Drug: Placebo Oral Tablet
- HL237 800mg (Experimental): take oral tablet once
  Interventions: Drug: HL237; Drug: Placebo Oral Tablet
- HL237 1200mg (Experimental): take oral tablet once
  Interventions: Drug: HL237; Drug: Placebo Oral Tablet
- HL237 1600mg (Experimental): take oral tablet once
  Interventions: Drug: HL237; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: HL237 — Experimental
Drug: Placebo Oral Tablet — placebo with same properties except for active ingredient

SUMMARY:
HL237 is a new autoimmune therapeutic agent for rheumatoid arthritis, including the basic structure of biguanide in metformin, an existing diabetes drug.

The immune modulating activity of HL237 was demonstrated in animal model. HL237 is a STAT3 inhibitor and STAT3 is well known for an important regulator inhibiting Th17 cells and activating Treg cells.

Therefore, when STAT3 activity is inhibited, it is expected to be able to treat autoimmune diseases such as rheumatoid arthritis.

This is the first clinical trial to be conducted for the development of HL237 and this clinical trial is for determining the maximum oral dose of HL237 and assessing safety, tolerability, and pharmacokinetic characteristics for each dose group.

ELIGIBILITY:
Inclusion Criteria:

* A healthy adult male aged 20 years or older and 45 years old at the time of the screening test
* Those who weigh more than 55kg but weigh less than ± 20% of ideal body weight
* Proper contraception during the clinical trial period
* After hearing the detailed explanation of the clinical trial, those who decide to participate voluntarily and write agreement

Exclusion Criteria:

* Clinically significant, a person with a history of neurological, psychiatric, malignant, cardiovascular, respiratory, kidney, endocrine, hematologic, digestive or central disease
* a person with a history of gastrointestinal disorders that may affect the absorption of pharmaceuticals for clinical trials (Crohn's disease, ulcers, etc.) or gastrointestinal surgery (except for simple cecal surgery or hernia surgery)
* a person with a history of hypersensitivity or clinically significant hypersensitivity to the clinical trial drug or additives
* a person judged to be inappropriate for the subject by health screening (history of disease, physical examination, vital signs, electrocardiogram, laboratory test, etc.)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 3days after administration
  maximum serum concentration after the drug has been administrated
Area Under the Curve [AUC] | 3days after administration
half life [t1/2] | 3days after administration

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 14days after administration

CONTACTS AND LOCATIONS:
Locations (1):
- The catholic university of korea seoul ST. mary's hospital, Soeul, South Korea